CLINICAL TRIAL: NCT02281318
Title: A Randomised, Double-blind, Placebo-controlled, Parallel-group, Multi-centre 24-week Study to Evaluate the Efficacy and Safety of Mepolizumab Adjunctive Therapy in Subjects With Severe Eosinophilic Asthma on Markers of Asthma Control
Brief Title: Efficacy and Safety Study of Mepolizumab Adjunctive Therapy in Participants With Severe Eosinophilic Asthma on Markers of Asthma Control
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200862
Record Dates: First submitted 2014-10-30; First posted 2014-11-03 (Estimated); Results first posted 2017-05-04 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Asthma
Keywords: Asthma control; Lung function; Health-related quality of life; Mepolizumab; Severe Eosinophilic asthma
MeSH Terms: conditions — Asthma; Pulmonary Eosinophilia | interventions — mepolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mepolizumab SC (Experimental): Participants will receive Mepolizumab 100 mg subcutaneously (SC) into the upper arm or thigh every 4 weeks for a period of 24 weeks (total of 6 doses) along with their respective standard care of treatment
  Interventions: Biological: Mepolizumab; Drug: SOC
- Placebo SC (Placebo Comparator): Participants will receive placebo (0.9% sodium chloride) subcutaneously into the upper arm or thigh every 4 weeks for a period of 24 weeks (total of 6 doses) along with their respective standard care of treatment
  Interventions: Drug: Placebo; Drug: SOC

INTERVENTIONS:
Biological: Mepolizumab — Humanised Immunoglobulin G (IgG) antibody (IgG1, kappa) with human heavy and light chain frameworks, provided as a lyophilised cake in sterile vial. Vial to be reconstituted with sterile water for injection, just prior to use
  Arms: Mepolizumab SC
Drug: Placebo — Sterile 0.9% sodium chloride solution
  Arms: Placebo SC
Drug: SOC — Standard of Care (SOC) will differ by participants, however it will include high dose ICS with at least one other controller, e.g. LABA, with or without maintenance OCS

SUMMARY:
This is a multi-centre, placebo-controlled, double-blind, parallel-group study to evaluate the efficacy and safety of mepolizumab adjunctive therapy in participants with severe eosinophilic asthma on markers of asthma control. The overall intent of the current study is to more fully explore the impact of mepolizumab on health-related quality of life (HR-QoL) and other measures of asthma control, including lung function.

Participants who meet the predefined criteria will be randomised to receive either mepolizumab or placebo in addition to standard of care asthma treatment. Approximately 780 participants with severe eosinophilic asthma will be screened to ensure the randomisation of 544 participants (272 participants per treatment group) into the study.

ELIGIBILITY:
Inclusion Criteria:

* Age: At least 12 years of age at the time of signing the informed consent/assent (For those countries where local regulations permit enrolment of adults only, participant recruitment will be restricted to those who are >=18 years of age)
* Inhaled Corticosteroid: A well-documented requirement for regular treatment with high dose inhaled corticosteroid (ICS) in the 12 months prior to Visit 1 with or without maintenance oral corticosteroids (OCS). For participants >=18 years old: ICS dose must be >=880 micrograms (mcg)/day fluticasone propionate (FP) (exactuator) or equivalent daily. For ICS/long-acting beta-2-agonist (LABA) combination preparations, the highest approved maintenance dose in the local country will meet this ICS criterion. For participants >=12 to <=17 years old: ICS dose must be >=440 mcg/day FP (ex-actuator) or equivalent daily. For ICS/LABA combination preparations, the mid-strength approved maintenance dose in the local country will meet this ICS criterion
* Controller Medication: Current treatment with an additional controller medication, besides ICS, for at least 3 months or a documented failure in the past 12 months of an additional controller medication for at least 3 successive months (e.g. LABA, leukotriene receptor antagonist [LTRA], or theophylline)
* Eosinophilic asthma: Prior documentation of eosinophilic asthma or high likelihood of eosinophilic asthma as per Randomisation Criteria 1 and 2
* FEV1: Persistent airflow obstruction as indicated by : For participants >=18 years of age at visit 1, a pre-bronchodilator FEV1 <80% predicted (National Health and Nutrition Examination Survey [NHANES III]) recorded at Visit 1. For participants 12-17 years of age at Visit 1: A pre-bronchodilator FEV1 <90% predicted (NHANES III) recorded at Visit 1 OR FEV1:FVC ratio <0.8 recorded at Visit 1
* Exacerbation history: Previously confirmed history of two or more exacerbations requiring treatment with systemic Corticosteroid (CS) (intramuscular, intravenous, or oral), in the 12 months prior to visit 1, despite the use of high-dose inhaled corticosteroids (ICS). For participants receiving maintenance CS, the CS treatment for the exacerbations must have been a two-fold dose increase or greater.
* Gender: Male or Eligible Female. To be eligible for entry into the study, females of childbearing potential must commit to consistent and correct use of an acceptable method of birth control listed in the protocol for the duration of the trial and for 4 months after the last study drug administration.
* Informed Consent/Assent: Able to give written informed consent/assent prior to participation in the core study, which will include the ability to comply with the requirements and restrictions listed in the consent/assent form and in this protocol. Participants must be able to read, comprehend, and write at a level sufficient to complete study related materials. Written informed consent must be obtained from ALL patients/legally authorized representative(s); for patients 12-17 years old, written informed assent must be obtained in addition to the legally authorized representative(s)' consent.
* French participants: In France, a participant will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

Exclusion Criteria:

* Smoking history: Current smokers or former smokers with a smoking history of >=10 pack years (number of pack years = (number of cigarettes per day/20) x number of years smoked). A former smoker is defined as a participant who quit smoking at least 6 months prior to Visit 1.
* Concurrent Respiratory Disease: Presence of a known pre-existing, clinically important lung condition other than asthma. This includes current infection, bronchiectasis, pulmonary fibrosis, bronchopulmonary aspergillosis, or diagnoses of emphysema or chronic bronchitis (chronic obstructive pulmonary disease other than asthma) or a history of lung cancer.
* Malignancy: A current malignancy or previous history of cancer in remission for less than 12 months prior to screening (Participants that had localized carcinoma of the skin which was resected for cure will not be excluded).
* Liver Disease: Known, pre-existing, unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, esophageal or gastric varices or persistent jaundice), cirrhosis, and known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Cardiovascular: Participants who have severe or clinically significant cardiovascular disease uncontrolled with standard treatment. Including but not limited to: (a) known ejection fraction of <30% OR (b) severe heart failure meeting New York Heart Association Class IV classification OR (c) hospitalised in the 12 months prior to Visit 1 for severe heart failure meeting New York Heart Association Class III OR (d) angina diagnosed less than 3 months prior to Visit 1 or at Visit 1.
* Other Concurrent Medical Conditions: Participants who have known, pre-existing, clinically significant endocrine, autoimmune, metabolic, neurological, renal, gastrointestinal, hepatic, haematological or any other system abnormalities that are uncontrolled with standard treatment.
* Eosinophilic Diseases: Participants with other conditions that could lead to elevated eosinophils such as Hypereosinophilic Syndromes, including Churg-Strauss Syndrome (Eosinophilic Granulomatosis with Polyangiitis [EGPA]), or Eosinophilic Esophagitis. Participants with a known, pre-existing parasitic infestation within 6 months prior to Visit 1 are also to be excluded.
* Electrocardiogram (ECG) Assessment: QT interval corrected for heart rate by Fridericia's formula (QTc(F)) >=450 milliseconds (msec) or QTc(F) >=480 msec for participants with Bundle Branch Block at Visit 1.
* Alcohol/Substance Abuse: A history (or suspected history) of alcohol misuse or substance abuse within 2 years prior to Visit 1.
* Immunodeficiency: A known immunodeficiency (e.g. human immunodeficiency virus [HIV]), other than that explained by the use of corticosteroids taken as therapy for asthma.
* Xolair: Participants who have received omalizumab (Xolair) within 130 days of Visit 1.
* Other Monoclonal Antibodies: Participants who have received any monoclonal antibody (other than Xolair) to treat inflammatory disease within 5 half-lives of Visit 1.
* Investigational Medications: Participants who have received treatment with an investigational drug within the past 30 days or five terminal phase half-lives of the drug whichever is longer, prior to Visit 1 (this also includes investigational formulations of marketed products).
* Hypersensitivity: Participants with allergy/intolerance to a monoclonal antibody or biologic.
* Pregnancy: Participants who are pregnant or breastfeeding. Patients should not be enrolled if they plan to become pregnant during the time of study participation. A urine pregnancy test is required of all women of child bearing potential. This test will be performed at the time points specified in the Time and Events Schedule in protocol.
* Adherence: Participants who have known evidence of lack of adherence to controller medications and/or ability to follow physician's recommendations.
* Previous participation: Previously participated in any study with mepolizumab and received investigational product (including placebo)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 556 (Actual)
Dates: Start 2014-12-11 (Actual); Primary Completion 2016-06-10 (Actual); Study Completion 2016-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (129):
- United States (23):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Rolling Hills Estates, California
  - GSK Investigational Site, Upland, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Gastonia, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Upland, Pennsylvania
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Rapid City, South Dakota
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Williamsburg, Virginia
- Argentina (7):
  - GSK Investigational Site, La Plata, Buenos Aires
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, Concepción del Uruguay, Entre Ríos Province
  - GSK Investigational Site, San Rafael, Mendoza Province
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Mendoza
- Belgium (5):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Erpent
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège
- Bulgaria (2):
  - GSK Investigational Site, Pleven
  - GSK Investigational Site, Sofia
- Canada (10):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Burlington, Ontario
  - GSK Investigational Site, St-Charles-Borromée, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Windsor, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Sainte-Foy, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec
- Czechia (7):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Hlučín
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Kralupy nad Vltavou
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Pilsen
  - GSK Investigational Site, Prague
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- France (10):
  - GSK Investigational Site, Brest
  - GSK Investigational Site, Dijon
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pessac
  - GSK Investigational Site, Reims
- Germany (8):
  - GSK Investigational Site, Bamberg, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Witten, North Rhine-Westphalia
  - GSK Investigational Site, Koblenz, Rhineland-Palatinate
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Schleswig, Schleswig-Holstein
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Greece (4):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Haidari / Athens
  - GSK Investigational Site, Rethymnon, Crete
  - GSK Investigational Site, Thessaloniki
- Italy (7):
  - GSK Investigational Site, Chieti, Abruzzo
  - GSK Investigational Site, Bari, Apulia
  - GSK Investigational Site, Foggia, Apulia
  - GSK Investigational Site, Parma, Emilia-Romagna
  - GSK Investigational Site, Reggio Emilia, Emilia-Romagna
  - GSK Investigational Site, Florence, Tuscany
  - GSK Investigational Site, Pisa, Tuscany
- Netherlands (5):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Leeuwarden
  - GSK Investigational Site, Leiden
  - GSK Investigational Site, Rotterdam
- Norway (4):
  - GSK Investigational Site, Bergen
  - GSK Investigational Site, Oslo
  - GSK Investigational Site, Stavanger
  - GSK Investigational Site, Trondheim
- Peru (4):
  - GSK Investigational Site, Lima, Lima Province
  - GSK Investigational Site, San Martín de Porres, Lima region
  - GSK Investigational Site, San Miguel, Lima region
  - GSK Investigational Site, Lima
- Russia (9):
  - GSK Investigational Site, Irkutsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saint Petesburg
  - GSK Investigational Site, Sestroretsk
  - GSK Investigational Site, Stavropol
  - GSK Investigational Site, Voronezh
  - GSK Investigational Site, Yekaterinburg
- Slovakia (4):
  - GSK Investigational Site, Bojnice
  - GSK Investigational Site, Spišská Nová Ves
  - GSK Investigational Site, Šaľa
  - GSK Investigational Site, Vráble
- Spain (8):
  - GSK Investigational Site, Alcorcón (Madrid)
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Pozuelo de Alarcón/Madrid
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Valencia
- Ukraine (6):
  - GSK Investigational Site, Dnipro
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Odesa
  - GSK Investigational Site, Vinnytsia
  - GSK Investigational Site, Zaporizhia
- United Kingdom (4):
  - GSK Investigational Site, Bradford
  - GSK Investigational Site, Oxford
  - GSK Investigational Site, Plymouth
  - GSK Investigational Site, Swansea

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Lemiere C, Taille C, Lee JK, Smith SG, Mallett S, Albers FC, Bradford ES, Yancey SW, Liu MC. Impact of baseline clinical asthma characteristics on the response to mepolizumab: a post hoc meta-analysis of two Phase III trials. Respir Res. 2021 Jun 22;22(1):184. doi: 10.1186/s12931-021-01767-z. PMID 34158028
- [Derived] Gibson PG, Prazma CM, Chupp GL, Bradford ES, Forshag M, Mallett SA, Yancey SW, Smith SG, Bel EH. Mepolizumab improves clinical outcomes in patients with severe asthma and comorbid conditions. Respir Res. 2021 Jun 7;22(1):171. doi: 10.1186/s12931-021-01746-4. PMID 34098955
- [Derived] Yancey SW, Ortega HG, Keene ON, Bradford ES. Efficacy of add-on mepolizumab in adolescents with severe eosinophilic asthma. Allergy Asthma Clin Immunol. 2019 Sep 3;15:53. doi: 10.1186/s13223-019-0366-x. eCollection 2019. PMID 31507641
- [Derived] Nelsen LM, Cockle SM, Gunsoy NB, Jones P, Albers FC, Bradford ES, Mullerova H. Impact of exacerbations on St George's Respiratory Questionnaire score in patients with severe asthma: post hoc analyses of two clinical trials and an observational study. J Asthma. 2020 Sep;57(9):1006-1016. doi: 10.1080/02770903.2019.1630640. Epub 2019 Jun 28. PMID 31251094
- [Derived] Yancey SW, Bradford ES, Keene ON. Disease burden and efficacy of mepolizumab in patients with severe asthma and blood eosinophil counts of >/=150-300 cells/muL. Respir Med. 2019 May;151:139-141. doi: 10.1016/j.rmed.2019.04.008. Epub 2019 Apr 8. PMID 31047111
- [Derived] Ortega H, Menzies-Gow A, Llanos JP, Forshag M, Albers F, Gunsoy N, Bradford ES, Yancey SW, Kraft M. Rapid and Consistent Improvements in Morning PEF in Patients with Severe Eosinophilic Asthma Treated with Mepolizumab. Adv Ther. 2018 Jul;35(7):1059-1068. doi: 10.1007/s12325-018-0727-8. Epub 2018 Jun 15. PMID 29949045
- [Derived] Chupp GL, Bradford ES, Albers FC, Bratton DJ, Wang-Jairaj J, Nelsen LM, Trevor JL, Magnan A, Ten Brinke A. Efficacy of mepolizumab add-on therapy on health-related quality of life and markers of asthma control in severe eosinophilic asthma (MUSCA): a randomised, double-blind, placebo-controlled, parallel-group, multicentre, phase 3b trial. Lancet Respir Med. 2017 May;5(5):390-400. doi: 10.1016/S2213-2600(17)30125-X. Epub 2017 Apr 5. PMID 28395936
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 200862 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 200862 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 200862 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 200862 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 200862 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 200862 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 200862 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 830 participants (par.) were screened (Visit 1) and entered into the run-in period, of which 556 participants were randomized and 551 participants received either mepolizumab 100 milligrams (mg) or placebo in addition to standard of care asthma treatment.
Groups:
- Placebo: Participants received placebo subcutaneously in upper arm or thigh following randomization at Visit 2 (Week 0) and every 4 weeks thereafter (last dose at Week 20) along with their standard of care asthma treatment up to 24 weeks.
- Mepolizumab 100 mg: Participants received mepolizumab 100 mg subcutaneously in upper arm or thigh following randomization at Visit 2 (Week 0) and every 4 weeks thereafter (last dose at Week 20) along with their standard of care asthma treatment up to 24 weeks.
Period: Overall Study
Arm/Group | Placebo | Mepolizumab 100 mg
Started | 277 | 274
Completed | 263 | 269
Not Completed | 14 | 5
Not completed — Adverse Event | 2 | 2
Not completed — Lack of Efficacy | 2 | 0
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Mepolizumab 100 mg | Total
Number analyzed (Participants) | 277 | 274 | 551
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.1 (12.94) | 49.8 (14.01) | 51.0 (13.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 176 | 149 | 325
  Male | 101 | 125 | 226
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 10 | 9 | 19
  Asian-Central/South Asian Heritage | 0 | 1 | 1
  Asian-East Asian Heritage | 0 | 2 | 2
  Asian-South East Asian Heritage | 0 | 1 | 1
  Black or African American | 7 | 8 | 15
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  White-Arabic/North African Heritage | 8 | 1 | 9
  White-White/Caucasian/European Heritage | 251 | 251 | 502

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline (BL) in St. George's Respiratory Questionnaire (SGRQ) Score at Week 24
Description: SGRQ consisted of 50 questions (scored from 0 to 100 where 0 indicates best and 100 indicates worst health) designed to measure Quality of Life in par. with diseases of airway obstruction, measuring symptoms, impact, and activity. Questions were completed by the par. with a recall over the past 4 weeks. SGRQ Total Score was calculated by summing the pre-assigned weights of answers, dividing by the sum of the maximum weights for items in SGRQ and multiplying by 100 to get a %. Change from BL in SGRQ was calculated as value at Week 24 minus value at BL for each par. and was analyzed using mixed model repeated measures allowing for covariates of BL value, region, BL maintenance oral corticosteroid (OCS) therapy, exacerbations in the year prior to the study (as an ordinal variable), BL % predicted FEV1 and visit, plus interaction terms for visit by BL and visit by treatment group. Modified Intent-to-Treat (mITT) Population consisted of all randomized par. who received >= 1 dose of drug.
Time Frame: Baseline and Week 24
Population: mITT Population. Participants with a missing Baseline covariate value or with no observed change from Baseline at any time point were excluded from the analysis model.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Mepolizumab 100 mg
Number analyzed (Participants) | 260 | 265
Scores on a scale | -7.9 (1.01) | -15.6 (1.00)
Statistical Analysis 1: Comparison: Placebo vs Mepolizumab 100 mg; Test type: Superiority or Other; p < 0.001, Mixed model repeated measures analysis; Mean Difference (Final Values) = -7.7, 95% CI 2-sided [-10.5 to -4.9]

2. Secondary Outcome: Mean Change From Baseline in Clinic Pre-bronchodilator Forced Expiratory Volume in One Second (FEV1) at Week 24
Description: FEV1 is the volume of air that can be forced out in one second after taking a deep breath. The change from Baseline in pre-bronchodilator FEV1 was calculated as the value at Week 24 minus the value at Baseline for each subject and was analyzed using a mixed model repeated measures adjusting for Baseline absolute pre-bronchodilator FEV1, region, Baseline maintenance OCS therapy, exacerbations in the year prior to the study and visit, plus interaction terms for visit by Baseline and visit by treatment group.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Milliliters (mL)
Arm/Group | Placebo | Mepolizumab 100 mg
Number analyzed (Participants) | 259 | 264
Milliliters (mL) | 56 (26.2) | 176 (26.1)
Statistical Analysis 1: Comparison: Placebo vs Mepolizumab 100 mg; Test type: Superiority or Other; p = 0.001, Mixed model repeated measures analysis; Mean Difference (Final Values) = 120, 95% CI 2-sided [47 to 192]

3. Secondary Outcome: Percentage of Participants Achieving a 4 Point or Greater Reduction From Baseline in SGRQ Score at Week 24
Description: The percentage of participants achieving a 4 point or greater reduction from Baseline in SGRQ (scored from 0-100 with lower scores indicating better outcome) at Week 24 was compared between treatment groups using a logistic regression model with covariates of Baseline value, region, Baseline maintenance OCS therapy, exacerbations in the year prior to the study (as an ordinal variable) and Baseline % predicted FEV1.
Time Frame: Baseline (Visit 2-latest pre-dose assessment) and Week 24
Population: mITT Population. Participants with a missing Baseline covariate value were excluded from the analysis model.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Mepolizumab 100 mg
Number analyzed (Participants) | 275 | 273
Percentage of participants | 55 | 73
Statistical Analysis 1: Comparison: Placebo vs Mepolizumab 100 mg; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.23, 95% CI 2-sided [1.55 to 3.22]

4. Secondary Outcome: Mean Change From Baseline in Asthma Control Questionnaire (ACQ-5) Score at Week 24
Description: The ACQ-5 is a five-item questionnaire, designed to be self-completed by the participants. ACQ-5 score is the mean score of 5 questions, each assessed on a 0-6 point scale to give a mean ranging between 0-6 with lower scores indicating better outcome. The five questions inquired about the frequency and/or severity of symptoms over the previous week. The response options for all these questions consisted of a zero (no impairment/limitation) to six (total impairment/limitation) scale. The mean change from Baseline was calculated as the value at Week 24 minus the Baseline value for each participant and analyzed using a mixed model repeated measures allowing for covariates of Baseline value, region, Baseline maintenance OCS therapy, exacerbations in the year prior to the study (as an ordinal variable), Baseline % predicted FEV1 and visit, plus interaction terms for visit by Baseline and visit by treatment group.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Mepolizumab 100 mg
Number analyzed (Participants) | 261 | 266
Scores on a scale | -0.40 (0.064) | -0.80 (0.064)
Statistical Analysis 1: Comparison: Placebo vs Mepolizumab 100 mg; Test type: Superiority or Other; p < 0.001, Mixed model repeated measures analysis; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-0.58 to -0.22]

ADVERSE EVENTS:
Time Frame: All serious adverse events (SAEs) and on-treatment non-serious adverse events (AEs) were collected from the start of investigational product and until 28 days after the IP stop date (on-treatment) and to the end of the study for SAEs (Week 24).
Description: The Safety Population consisted of all randomized participants who received at least one dose of trial medication. Subjects were analysed according to treatment actually received.
Groups:
- Mepolizumab 100 mg SC: Participants received mepolizumab 100 mg subcutaneously in upper arm or thigh following randomization at Visit 2 (Week 0) and every 4 weeks thereafter (last dose at Week 20) along with their standard of care asthma treatment up to 24 weeks.
Arm/Group | Placebo | Mepolizumab 100 mg SC
Serious Adverse Events (participants affected / at risk) | 23/278 | 15/273
Other Adverse Events (participants affected / at risk) | 140/278 | 124/273
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=278) | Mepolizumab 100 mg SC (N=273)
Asthma (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Bronchitis bacterial (Infections and infestations) | 1 | 0
Catheter site infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Gastroenteritis rotavirus (Infections and infestations) | 1 | 0
Hemophilus infection (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 0 | 1
Localized infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Staphylococcal bacteremia (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 2 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 0 | 1
Vasculitis (Vascular disorders) | 1 | 0
Myocardial ischemia (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Allergic granulomatous angiitis (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Blood glucose increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=278) | Mepolizumab 100 mg SC (N=273)
Nasopharyngitis (Infections and infestations) | 46 | 31
Upper respiratory tract infection (Infections and infestations) | 14 | 17
Sinusitis (Infections and infestations) | 12 | 11
Bronchitis (Infections and infestations) | 11 | 6
Rhinitis (Infections and infestations) | 7 | 10
Headache (Nervous system disorders) | 59 | 45
Back pain (Musculoskeletal and connective tissue disorders) | 18 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 9
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 14 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 11
Fatigue (General disorders) | 11 | 7
Nausea (Gastrointestinal disorders) | 7 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.